CLINICAL TRIAL: NCT04495426
Title: Genetic Mechanism of Conserved Ancestral Haplotype in SCA10
Acronym: CAHSCA10
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Tetsuo Ashizawa, MD, Neurosciences Research Program, Director, The Methodist Hospital Research Institute
Other Study IDs: Pro00022772
Record Dates: First submitted 2020-07-13; First posted 2020-07-31 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Spinocerebellar Ataxia Type 10
Keywords: SCA10; genotype; spinocerebellar; ataxia; type 10; cerebellum; G allele; haplotype
MeSH Terms: conditions — Spinocerebellar Ataxia 10; Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be stored with new ID for de-identification and used for DNA analysis and RNA repository. Sperm samples will be obtained by ejaculating semen into a condom or directly into a urine specimen collection container during a sexual activity.
  A subset of symptomatic (up to 5) and at-risk individuals (up to 10) will be invited to a follow-up visit to collect a skin biopsy. PIs will choose candidates for this invitation, based on their SCA10 haplotypes and type of expansions. In order to preserve genetic status blinding of at-risk subjects, for each premanifest carrier chosen, a non-carrier will be also invited to be a donor of a skin biopsy. A fibroblast culture will be established and stored in a bio-repository for further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Presence of symptomatic ataxic disease: Presence of symptomatic ataxic disease with definite molecular diagnosis of SCA10 or whose first-degree relative has a molecular diagnosis of SCA10.
  Interventions: Other: Non-interventional study
- Premanifest for SCA10: Asymptomatic participants of either sex aged ≥18 with definite molecular diagnosis of SCA10 (Premanifest carriers)
  Interventions: Other: Non-interventional study
- At risk for SCA10: Asymptomatic participants of either sex, aged ≥18 whose first-degree relative has a molecular diagnosis of SCA10 (50%-at-risk relatives*).
  Interventions: Other: Non-interventional study
- Non-carrier for SCA10 (Control): At risk participants who test negative for the SCA10 mutation will serve as non-carriers. Exclusion criteria described above also applies to non-carrier subjects. If the number of non-carriers were less than 10, we will recruit additional participants from normal population to supplement the controls.
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — There are no treatments to stop or even slow down the progression of this disease although there are treatments that temporarily improve the symptoms, such as anti-seizure medications.

SUMMARY:
Spinocerebellar ataxia type 10 (SCA10) is a hereditary ataxia whose ancestral mutation occurred in East Asia. The mutation is likely to have migrated during peopling of American continents from East Asia. We found a specific rare DNA variation associated with SCA10. We test whether this variation played a key role in the birth and subsequent spreading of SCA10 mutation.

DETAILED DESCRIPTION:
Spinocerebellar ataxia type 10 (SCA10) is a rare ataxic disorder due to a large expansion of intronic (ATTCT)n repeat in ATXN10. SCA10 afflicts primarily Latin American (LA) populations of Native American Ancestry; recent discoveries of two East Asian (EA) SCA10 families suggests an Asian origin. SCA10 families from LA and EA share an ancestral haplotype that includes the G allele (allele frequency: 2-4% in EA and LA populations but 0% elsewhere) of a C/G/T single nucleotide polymorphism (SNP) at rs41524745 (https://www.ncbi.nlm.nih.gov/snp/rs41524547#frequency_tab). Two characteristics suggest that rs41524745 has a functional role over the expansion: this SNP resides in the sequence encoding miR4762; and total linkage between the SNP and the SCA10 repeat, although they are ~35kb apart, a distance sufficient for multiple recombination events within the 15,000-20,000 years since human migration across Bering landmass. We studied DNA samples with G allele at rs41524547 from the 1000 Genomes repository and our own samples from general populations and surprisingly found 0-25% of these G(+) samples have SCA10 repeat expansions. Since our genotype-phenotype data suggest that SCA10 expansions with (ATTCC)n or (ATCCT)n(ATCCC)n repeat insertion in the 3' end of (ATTCT)n expansion exhibit full penetrance while pure (ATTCT)n expansion has reduced penetrance, the last one can be more common than previously expected. Hypotheses: (1) the G allele at rs41524547 predisposes the SCA10 (ATTCT)n repeat for expansion (Type A expansion), that remains mostly non-penetrant, and (2) the (ATTCT)n-(ATTCC)n (Type B) or (ATTCT)n(ATCCT)n-(ATCCC)n (Type C) repeat drives the SCA10 pathogenicity. To test the hypothesis, we propose three Aims in close collaborations between US and Brazilian SCA10 consortia:

Aim 1. To determine the relationship between SCA10 and the G allele at rs41524547.

Aim 2. To confirm that Type B and Type C expansions are pathogenic, but Type A expansions have significantly reduced pathogenicity.

Aim 3. To determine if the G allele at rs41524547 reduces downstream recombination rates, protects against the toxicity of SCA10 RNA expansions, or promote expanded states of the SCA10 repeat.

This effort will enable long term goals to: (1) identify people at risk for SCA10 by high-throughput screening of general populations for the G allele at rs41524547 in Brazil, (2) determine the frequency of non-penetrant SCA10 expansion alleles in Brazil, and (3) develop treatments of SCA10 based on results of this project.

The proposed project requires complimentary expertise in multiple areas, including coordination of the clinical studies, along with recruitment plans and executions, management of tissue repository, maintenance and expansion of the clinical database, clinical MR technology and data analyses, which will be ongoing in both the US and Brazil.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (no study-related procedures may be performed before the subject has signed the consent form).
2. Participants of either sex aged ≥18 with presence of symptomatic ataxic disease with definite molecular diagnosis of SCA10 or whose first-degree relative has a molecular diagnosis of SCA10.
3. Asymptomatic participants of either sex aged ≥18 with definite molecular diagnosis of SCA10 (Premanifest carriers) or those whose first-degree relative has a molecular diagnosis of SCA10 (50%-at-risk relatives*).
4. Participants capable of understanding and complying with protocol requirements.

Exclusion Criteria:

1. Known genotype consistent with other inherited ataxias.
2. Concomitant disorder(s) or condition(s) that affects assessment of ataxia or severity of ataxia during this study.
3. Unwillingness to provide a DNA sample at study entry.
4. Inability to undergo MRI scanning, Weight over 300lbs, Presence of structural abnormalities such as subdural hematoma or primary or metastatic neoplasms, concurrent illnesses or treatment interfering with cognitive function such as stroke or normal pressure hydrocephalus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit symptomatic participants, premanifest carriers and related non-carriers (at-risk siblings without a SCA10 expansion) members of SCA10 families who have been diagnosed with Spinocerebellar ataxia type 10 (SCA10) or those whose first-degree relative has a molecular diagnosis or SCA10.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Examine the disease progression in SCA10 as determined by change in the scale for the assessment and rating of ataxia score compared to healthy controls | Baseline visit 1, Follow up visit (12-18 months after visit 1)
  Scale for the assessment and rating of ataxia (SARA) was evaluated in two large validation trials performed by the EUROSCA clinical group and was found to be easy to use, reliable and valid. SARA has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
Examine the disease progression in SCA10 as determined by change in Spinocerebellar Ataxia Functional Index score compared to healthy controls | Baseline visit 1, Follow up visit (12-18 months after visit 1)
  The Spinocerebellar Ataxia Functional Index (SCAFI) is composed of:
  1. Timed 8 meter walk at maximum speed (8MW). Times are only given for two successfully completed trials. Discontinue the test if participant cannot complete trial in 3 minutes (more severe ataxia).
  2. Timed dexterity test: 9-hole peg test (9HPT). Times are only given for two successfully completed trials for each hand. If participant cannot complete one trial in 5 minutes (more severe ataxia) discontinue 9-hole-peg test.
  3. Timed speech test: PATA rate, a measure of speech performance. The participant is asked to repeat "PATA" as quickly and distinctly as possible for 10 seconds until told to stop. As soon as the participant begins speaking, start timer and begin counting the number of PATA repeats. Higher number (less dysarthria), lower number (more dysarthria). Discontinue if PATA articulation is too difficult to distinguish for counting or if participant cannot complete 10 seconds for two consecutive trials.
Examine the disease progression in SCA10 as determined by change in Composite Cerebellar Functional Severity Score compared to healthy controls | Baseline visit 1, Follow up visit (12-18 months after visit 1)
  The Composite Cerebellar Functional Severity (CCFS) score is a quantitative tool to measure cerebellar severity independently from age. It is an assessment in addition to a clinical examination and has demonstrated its usefulness in epidemiological studies, clinical trials, and patient follow-up that only take 5 minutes to be administrated. The CCFS is a combination of the time to perform 2 tasks; a 9-hole pegboard and a click test. It was validated in adults and children. CCFS scores range from 0.50 (normal/no ataxia) to 1.80 (more severe ataxia).
Examine the disease progression in SCA10 as determined by change in Neurological Examination Score for Spinocerebellar Ataxia compared to healthy controls | Baseline visit 1, Follow up visit (12-18 months after visit 1)
  The Neurological Examination Score for Spinocerebellar Ataxia (NESSCA) scale is based on the standardized neurological examination, and consists of 18 items that yield a total score ranging from 0 (no ataxia) to 40 (most severe ataxia). The NESSCA is a comprehensive measure of disease severity that was shown to be both clinically useful and scientifically valid.
Examine the disease progression in SCA10 as determined by change in Inventory of Non-ataxia Symptoms score compared to healthy controls | Baseline visit 1, Follow up visit (12-18 months after visit 1)
  The Inventory of Non-ataxia Symptoms (INAS) is a scale utilized in recording the occurrence of accompanying non-ataxia symptoms. In the SARA validation trials, INAS was applied to a large number of SCA patients. For a semiquantitative assessment of non-ataxia signs, the number of non-ataxia signs is counted yielding the INAS count, a dimensionless value with a range from 0 (no ataxia) to 16 (most severe ataxia). To determine the INAS count, only the presence or absence of one of the 16 signs is considered. Statistical evaluation showed good reliability.
Examine the disease progression in SCA10 as determined by change in Beck Depression Inventory score compared to healthy controls | Baseline visit 1, Follow up visit (12-18 months after visit 1)
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Answers can range from 0 to 3 for each item. The total score will range from 0 (considered normal) to 40 (extreme depression).
Examine the disease progression in SCA10 as determined by change in Europe Quality of Life-5 Dimension score compared to healthy controls | Baseline visit 1, Follow up visit (12-18 months after visit 1)
  The Europe Quality of Life-5 Dimension (Euro Qol-5D or EQ-5D), is a measure developed by the EuroQol Group that generates a single index value for health status with considerable potential for use in health care evaluation.The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Number of participants with Electroencephalography changes that may be distinctive for SCA10 | Baseline visit 2 (within 6 weeks of visit 1)
  Electroencephalography (EEG) will be obtained and analyzed for changes that may be distinctive for SCA10: seizure spikes and/or sharp waves during and, sometimes, between seizure episodes.
Examine the level of disease activity based on change in cerebellar and brainstem volumes compared to healthy controls | Baseline visit 2 (within 6 weeks of visit 1)
  Magnetic Resonance Imaging (MRI) using a 3T scanner will be used to measure cerebellar and brainstem volumes.
Examine the level of disease activity based on change in grey matter and white matter loss metrics from voxel-based morphometry compared to healthy controls | Baseline visit 2 (within 6 weeks of visit 1)
  Magnetic Resonance Imaging (MRI) will be used to measure change in grey matter volume and white matter volume from voxel-based morphometric data.
Examine the level of disease activity based on change in mean diffusivity compared to healthy controls | Baseline visit 2 (within 6 weeks of visit 1)
  Magnetic Resonance Imaging (MRI) will be used to measure change in mean diffusivity.
Examine the level of disease activity based on change in radial and axial diffusivity compared to healthy controls | Baseline visit 2 (within 6 weeks of visit 1)
  Magnetic Resonance Imaging (MRI) will be used to measure change in radial and axial diffusivity.

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuo A, MD, Principal Investigator — National Institute of Neurological Diseases
Locations (3):
- Houston Methodist Hospital, Houston, Texas, United States
- Brazil (2):
  - Universidade Federal do Paraná, Paraná, Curibita
  - Hospital de Clinicas de Porto Alegre, Porto Alegre